CLINICAL TRIAL: NCT04322383
Title: Phase 2 Trial for Binimetinib for Patients With Relapsed/Refractory BRAF Wild Type Hairy Cell Leukemia and Variant
Brief Title: Binimetinib for People With Relapsed/Refractory BRAF Wild Type Hairy Cell Leukemia and Variant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200075; 20-C-0075
Record Dates: First submitted 2020-03-25; First posted 2020-03-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08-22

CONDITIONS: Hairy Cell Leukemia
Keywords: MEK1; Inhibitor; MEK2; MEK162
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — binimetinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1/Experimental therapy (Experimental): Treatment with binimetinib
  Interventions: Drug: binimetinib

INTERVENTIONS:
Drug: binimetinib — Binimetinib will be given orally at a dose of 45mg BID continuously for 28-day cycles with no resting period between cycles.

SUMMARY:
Background:

Most people with hairy cell leukemia have a BRAF gene mutation. They can be treated with BRAF inhibitors, drugs that target this mutation. For people who do not have this mutation, BRAF inhibitors are not a treatment option. We found that in hairy cell leukemia, when BRAF is not mutated, the MEK gene frequently is. Binimetinib is a MEK inhibitor which targets MEK. It is important to determine if this drug can be a good treatment option in those who cannot benefit treatment with BRAF inhibitors.

Objective:

To see if binimetinib is an effective treatment for hairy cell leukemia that does not have a BRAF mutation.

Eligibility:

People ages 18 and older with hairy cell leukemia without a mutation in the BRAF gene and whose disease either did not respond to treatment or came back after treatment

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests
* Lung and heart tests
* Eye exam
* Bone marrow biopsy: A needle will be injected through the participant s skin into the bone to remove a sample of marrow.
* CT or MRI scan: Participants will lie in a machine that takes pictures of the body. They might receive a contrast agent by vein.

Before they start treatment, participants will have an abdominal ultrasound, pulmonary function tests, and exercise stress tests.

Participants will take binimetinib by mouth twice daily in 28-day cycles. They will keep a medication diary.

Participants will have at least one visit before every cycle. Visits will include repeats of some screening tests.

Participants may continue treatment as long as their disease does not get worse and they do not have bad side effects.

About a month after their last dose of treatment, participants will have a follow-up visit. They will then have visits once a year....

DETAILED DESCRIPTION:
Background:

* Hairy cell leukemia (HCL) is an indolent B-cell leukemia comprising 2 percent of all leukemias, or approximately 1300 new cases per year in the US.
* BRAF V600E mutation is very common in classic HCL.
* HCL variant (HCLv) is wild type for BRAF and is more aggressive compared to classic HCL due to its lower response and shorter duration of response to standard purine analog chemotherapy. The median survival is only ~6 years compared to >25 years for classic HCL.
* CD25+ classic-appearing HCL-cells that express unmutated IGHV4-34+ immunoglobulin rearrangement, are wild-type for BRAF, and confer a poor prognosis when treated with standard purine analog chemotherapy.
* While BRAF and MEK combination inhibition is making an impact in the treatment of BRAF V600E mutated HCL, this treatment is not applicable for patients with BRAF-WT HCL/HCLv. Furthermore, with poor survival outcomes in this patient population, lack of targeted therapy constitutes a clear unmet need.
* Recently, several BRAF WT HCL/HCLv patients have received MEK inhibitors by compassionate use and have had lifesaving partial to complete remission, however the response has not been assessed systematically in clinical trials.
* Binimetinib (also known as MEK162) is an orally bioavailable, selective and potent mitogenactivated protein (MAP) kinase (MEK1 and MEK2) inhibitor, which is approved for use in combination with encorafenib for the treatment of patients with BRAF-mutant melanoma
* We have described MAP2K1 (MEK) mutations which may drive the aggressive clinical behavior of BRAF WT HCL/HCLv patients, but MEK inhibition may be clinically useful even in these patients without known MAP2K1 (MEK) mutations.

Objective:

-To determine the overall response rate (ORR) to binimetinib, in participants with BRAF WT HCL and HCLv.

Eligibility:

* BRAF WT HCL or HCLv with at least 1 prior purine analog treatment
* Need for treatment as evidenced by any one of the following: ANC <1 x10^3/mcL, Hgb <10g/dL, Platelet count <100 x10^3/mcL, leukemia cell count >5 x10^3/mcL, symptomatic splenomegaly, enlarging HCL mass > 2cm in short axis.
* greater than or equal to 18 years of age.
* No uncontrolled infection, cardiopulmonary dysfunction, or secondary malignancy requiring treatment.
* No chemotherapy, immunotherapy, investigational agent or radiotherapy within 4 weeks prior to the start of study treatment.

Design:

* Single arm phase 2 trial to determine ORR in participants with relapsed/refractory BRAF WT HCL and HCLv.
* 2-phase minimax design will be used to rule out an unacceptable 10 percent in favor of an improved 25 percent ORR.
* Initially 16 evaluable participants will be enrolled. If 2 or more achieve a major response, then accrual will continue to a total of 31 evaluable participants.
* Binimetinib will be given at a dose of 45mg twice daily for as long as participants can continue dosing chronically without significant toxicity or a trial off therapy due to achievement of MRD negative complete remission or partial response (PR) / complete response (CR) in which they would like a trial off therapy. Participants may return to therapy within 2 years of stopping treatment if evidence of disease returns.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically confirmed diagnosis of HCL or HCLv according to morphological and immunophenotypic criteria of World Health Organization (WHO) classification [WHO, 2008 revised 2016] of lymphoid neoplasm. Participants should have at least one of the following indications for therapy:

  * Absolute neutrophil count (ANC) <1 x10^3/mcL
  * Hemoglobin <10g/dL
  * Platelets<100 x10^3/mcL
  * Symptomatic splenomegaly
  * Enlarging HCL mass or bone lesion > 2cm in short axis
  * Leukemia cell count >5x10^3/mcL
  * Leukemic doubling time <6 months

Participants who have eligible blood counts within 4 weeks prior to initiation of study therapy will not be considered ineligible if subsequent blood counts prior to initiation of study therapy fluctuate and become ineligible up until the time of the initiation of study therapy.

* Refractory or relapsed disease - defined as either:

  * Refractory- no response or disease progression in less than or equal to 1 year following first-line treatment with a purine analog, or
  * Relapsed- having relapsed following treatment with at least 1 prior purine-analog treatments
* Participants must be BRAF WT as confirmed from fresh bone marrow aspirate and/or peripheral blood sample, or lymph node/mass by the Laboratory of Pathology, NCI
* Participants who are ineligible for, unable to obtain in a timely manner, cannot access, unwilling to undergo or have failed Moxetumomab Pasudotox trial at NCI
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60 percent).
* Adequate organ and marrow function as defined below:

  * Total bilirubin less than or equal to 3x upper limit of normal (ULN), unless consistent with Gilbert s (ratio between total and direct bilirubin > 5)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3x ULN
  * Alkaline phosphatase <= 5x ULN
  * Serum creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal calculated using estimated glomerular filtration rate (eGFR)
  * Serum albumin greater than or equal to 2 g/dL
  * Prothrombin time (PT)/International Normalized Ratio (INR) < 2.5x ULN (If on warfarin, PT/INR < 3.5x ULN; If on any other anticoagulation, Prothrombin time (PT) < 2.5x ULN
  * Fibrinogen greater than or equal to 0.5x lower limit of normal
* The effects of binimetinib on the developing human fetus are unknown therefore participants must use effective methods of contraception as directed below.
* Females of childbearing potential (FOCBP) who are sexually active with a nonsterilized male partner must use a highly effective method of contraception and not donate ova prior to study entry and or the duration of study treatment and until 30 days after the last dose of binimetinib. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are premenarchal or postmenopausal (defined as 12 months with no menses without an alternative medical cause). A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Not all methods of contraception are highly effective. Female subjects must use a hormonal method in addition to a barrier method alone, to minimize the chance of pregnancy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Non-sterilized male participants who are sexually active with a female partner of childbearing potential must agree to use methods of contraception that are highly effective or acceptable, and not donate sperm from study entry until 90 days after the last dose of binimetinib.
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 3 days after the last dose of the study drug.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Must co-enroll in study 10-C-0066: Collection of Human Samples to Study Hairy Cell and other Leukemias, and to Develop Recombinant Immunotoxins for Cancer Treatment

EXCLUSION CRITERIA:

* Participants who have had chemotherapy, immunotherapy or radiotherapy within 2 weeks prior to the start of study treatment.
* Prior therapy with binimetinib.
* Participants who are receiving any other investigational agents or have received an investigational agent within 14 days prior to the start of study treatment.
* Participants who have undergone major surgery less than or equal to 6 weeks prior to start of study treatment or who have not recovered from side effects of such procedure.
* Known hypersensitivity or contraindication to any component of binimetinib or its excipients.
* Inability to swallow and retain study drug.
* Pregnant women as evaluated by a positive serum or urine beta-human chorionic gonadotropin (beta-hCG) test.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac disfunction (details as below), uncontrolled pulmonary infection, pulmonary edema or psychiatric illness/social situations that would limit compliance with study requirements.
* Evidence of active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection.

Note: Participants with laboratory evidence of cleared HBV or HCV infection may be enrolled. If positive for Hepatitis B core antibody or surface antigen, the participant must be on Tenofovir or Entecavir and Hepatitis B deoxyribonucleic acid (DNA) viral load (VL) must be <2000 IU/mL

* Active second malignancy requiring treatment other than minor resection of indolent cancers like basal cell and squamous skin cancers.
* Human immunodeficiency virus (HIV)-positive participants unless taking appropriate anti- HIV medications with a CD4 count of > 200. Otherwise, there may be an increased risk of infections.
* History of an allogeneic bone marrow or stem cell transplant.
* Impaired cardiovascular function or clinically significant cardiovascular disease including, but not limited to, any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 3 months prior to initiation of study therapy;
  * Congestive heart failure requiring treatment (New York Heart Association Grade greater than or equal to 2);
  * Left ventricular ejection fraction (LVEF) < 50 percent as determined by multigated acquisition scan (MUGA) or transthoracic echocardiogram (TTE);
  * Uncontrolled hypertension defined as persistent systolic blood pressure greater than or equal to 160 mmHg or diastolic blood pressure greater than or equal to 100 mmHg despite current therapy;
  * History or presence of clinically significant cardiac arrhythmias (including resting bradycardia, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * Triplicate average baseline QTcF interval greater than or equal to 480 ms.
* Impairment of gastrointestinal function or disease which may significantly alter the absorption of study drug (e.g., active ulcerative disease, uncontrolled vomiting or diarrhea, malabsorption syndrome, small bowel resection with decreased intestinal absorption), or recent (less than or equal to 3 months) history of a partial or complete bowel obstruction, or other conditions that will interfere significantly with the absorption of oral drugs.
* Concurrent neuromuscular disorder that is associated with elevated creatinine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of maculopathy or retinopathy for which there is an increased risk of

MEK induced exudation (e.g., Central Serous Retinopathy).

-History of thromboembolic or cerebrovascular events less than or equal to 12 weeks prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli.

Note: Participants with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks.

Note: Participants with thromboembolic events related to indwelling catheters or other procedures may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | every year
  Percentage of participants with the best overall response of CR or PR to therapy

SECONDARY OUTCOMES:
CR rate | every year
  the time criteria are met for CR or PR (whichever is recorded first) until the first date that participant no longer qualifies as a PR
Progression free survival | every year
  duration of time from the start of the treatment until time of disease relapse from PR, disease progression, or death, whichever occurs first
Overall survival | every year
  the time from the start of the treatment until time of death from any cause
time to next treatment | every year
  duration of time from the start of the binimetinib to next line of treatment
safety | every 4 weeks
  The fraction of participants with toxicity noted will be reported by grade and type of toxicity identified.
different response relative to MAP2K1 mutations | every year
  determine whether the response to binimetinib is different in participants with and without MAP2K1 (MEK mutations), in participants for which MEK status is known

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0075.html